CLINICAL TRIAL: NCT00431496
Title: A Study To Assess Achievement of NKF K/DOQI Targets Using Sensipar (Cinacalcet) in Australian Subjects With End Stage Renal Disease (ESRD) Who Are Being Treated With Aranesp for Anaemia Management
Brief Title: A Study of Cinacalcet to Improve Achievement of National Kidney Foundation Kidney Disease Outcomes Quality Initiative (K/DOQI) Targets in Patients With End Stage Renal Disease (ESRD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20040196; To Target
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Anemia; Secondary Hyperparathyroidism
Keywords: Anemia; Intact Parathyroid Hormone (iPTH); Secondary Hyperparathyroidism (SHPT)
MeSH Terms: conditions — Anemia; Hyperparathyroidism, Secondary | interventions — Cinacalcet

ARMS (1):
- Cinacalcet (Experimental): Cinacalcet was administered orally at a starting dose of 30 mg/day for 23 weeks. Possible sequential doses during the study were 30, 60, 90, 120, and 180 mg. Dose escalation of cinacalcet occurred if the intact parathyroid hormone (iPTH) level from the previous study visit was > 31.8 pmol/L (300 pg/mL) unless the participant had either reached the maximum dose (180 mg/day), the serum corrected total calcium was < 2.1 mmol/L (8.4 mg/dL), or the participant experienced an adverse event that precluded a dose increase.
  Interventions: Drug: Cinacalcet

INTERVENTIONS:
Drug: Cinacalcet — Cinacalcet tablets
  Other Names: Sensipar®

SUMMARY:
The purpose of this study is to show that the use of cinacalcet in patients with End Stage Renal Disease can help achieve NKF K/DOQI targets for both serum calcium and calcium phosphorous product.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD requiring maintenance dialysis (haemodialysis, haemodiafiltration, haemofiltration, or peritoneal dialysis) for at least 1 month
* Being treated with Aranesp for anaemia management and have stabilised haemoglobin (Hb) levels. Hb stabilisation is defined as two consecutive Hb measurements during the screening period (that must include the most recent assessment) above 110 g/L.
* Males or females > 18 years of age at the time of informed consent
* Patients participating in this study must agree to use, in the opinion of the principal investigator, highly effective contraceptive measures throughout the study. Females must have a negative serum pregnancy test within 21 days before day 1 if they are of child-bearing potential
* The mean of 2 Intact parathyroid hormone (iPTH) determinations within 21 days before study day 1 and drawn at least 2 days apart must be > 31.8 pmol/L (300 pg/mL) and < 84.8 pmol/L (800 pg/mL)
* The mean of 2 serum calcium determinations (corrected for albumin) drawn on the same day as the PTH determinations must be > 2.1 mmol/L (8.4 mg/dL)
* Signed the Independent Ethics Committee (IEC) approved Informed Consent document, before ANY study specific procedures are initiated

Exclusion Criteria:

* Have received vitamin D therapy for less than 21 days before day 1 or required a change in prescribed vitamin D brand or dose within 21 days before day 1. If patients are not prescribed vitamin D therapy, they must remain free of vitamin D therapy for the 21 days before day 1
* Have an unstable medical condition, defined as having been hospitalised, other than for dialysis vascular access revision, within 30 days before day 1, or otherwise unstable in the judgment of the investigator
* Hypersensitivity to Sensipar or any of its components
* Are currently breastfeeding
* Have had a parathyroidectomy in the 3 months before day 1
* Experienced a myocardial infarction within 3 months prior to day 1
* Have had a red blood cell transfusion within 3 months prior to day 1
* Are currently enrolled in, or have not yet completed at least 30 days before day 1 other invasive investigational device or investigational drug trials, or are receiving other investigational agents (experimental dialysis machines are acceptable)
* Have a gastrointestinal disorder that may be associated with impaired absorption of orally administered medications or an inability to swallow tablets
* Have a disorder that would interfere with understanding and giving informed consent, or compliance with protocol requirements
* Have previously enrolled in this study or participated in other trials of Sensipar

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 27 October 2006 through 31 December 2008
Groups:
- Cinacalcet: Cinacalcet was administered orally at a starting dose of 30 mg/day for 23 weeks. Possible sequential doses during the study were 30, 60, 90, 120, and 180 mg. Dose escalation of cinacalcet occurred if the intact parathyroid hormone (iPTH) level from the previous study visit was > 31.8 pmol/L (300 pg/mL), unless the participant had either reached the maximum dose (180 mg/day), the serum corrected total calcium was < 2.1 mmol/L (8.4 mg/dL), or the participant experienced an adverse event that precluded a dose increase.
Period: Overall Study
Arm/Group | Cinacalcet
Started | 71
Completed | 60
Not Completed | 11
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Protocol-specified criteria | 5

BASELINE CHARACTERISTICS:
Groups:
- Cinacalcet: Cinacalcet was administered orally at a starting dose of 30 mg/day for 23 weeks.
Arm/Group | Cinacalcet
Number analyzed (Participants) | 71
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.3 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 43
Race/Ethnicity, Customized [Number; unit: Participants]
  Aborigine | 3
  Asian | 6
  Black or African American | 1
  Native Hawaiian or Other Pacific Islander | 5
  White or Caucasian | 53
  Other | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Mean Intact Parathyroid Hormone Value Between 150 and 300 pg/mL and a Calcium - Phosphorus Product Value < 55 mg^2/dL^2
Description: The National Kidney Foundation Kidney Disease Outcomes Quality Initiative (NKF K/DOQI) recommends that treatment interventions to control parathyroid hormone should not result in significant elevation of calcium - phosphorus product (Ca x P; a derived value calculated from serum calcium and phosphorus levels). The primary objective of the study was to assess the simultaneous achievement of NKF K/DOQI targets of intact parathyroid hormone (iPTH) greater than or equal to 15.9 pmol/L and less than or equal to 31.8 pmol/L (150 - 300 pg/mL) and a Ca x P value < 4.44 mmol^2/L^2 (55 mg^2/dL^2) during the effectiveness assessment phase.
Time Frame: Weeks 17 to 23
Population: All participants who received cinacalcet
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 71
Participants | 30
Statistical Analysis 1: Comparison: Cinacalcet; Test type: Superiority or Other; Percentage of participants = 42.3, 95% CI [30.8 to 53.7]

2. Secondary Outcome: Number of Participants Who Achieved a Mean iPTH Value Between 150 and 300 pg/mL
Description: Number of participants who achieved a mean intact Parathyroid Hormone (iPTH) value greater than or equal to 15.9 and less than or equal to 31.8 pmol/L (150 - 300 pg/mL) during the effectiveness assessment phase.
Time Frame: Weeks 17 to 23
Population: All participants who received cinacalcet
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 71
Participants | 37
Statistical Analysis 1: Comparison: Cinacalcet; Test type: Superiority or Other; Percentage of participants = 52.1, 95% CI [40.5 to 63.7]

3. Secondary Outcome: Number of Participants Who Achieved a Mean Ca x P Value < 4.44 mmol^2/L^2 (55 mg^2/dL^2)
Description: The number of participants who achieved a mean serum calcium x phosphorus (Ca x P) value < 4.44 mmol^2/L^2 (55 mg^2/dL^2) during the effectiveness assessment phase. The calcium - phosphorus product is a derived value calculated from serum calcium and phosphorus levels.
Time Frame: Weeks 17 to 23
Population: All participants who received cinacalcet
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 71
Participants | 56
Statistical Analysis 1: Comparison: Cinacalcet; Test type: Superiority or Other; Percentage of participants = 78.9, 95% CI [69.4 to 88.4]

4. Secondary Outcome: Number of Participants Who Achieved a Mean Calcium Value ≥ 2.1 and ≤ 2.37 mmol/L
Description: The number of participants who achieved a mean corrected serum calcium (Ca) value ≥ 2.1 and ≤ 2.37 mmol/L (8.4 to 9.5 mg/dL) during the effectiveness assessment phase.
Time Frame: Weeks 17 to 23
Population: All participants who received cinacalcet
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 71
Participants | 39
Statistical Analysis 1: Comparison: Cinacalcet; Test type: Superiority or Other; Percentage of participants = 54.9, 95% CI [43.4 to 66.5]

5. Secondary Outcome: Number of Participants Who Achieved a Mean Phosphorus Value ≥ 1.13 and ≤ 1.78 mmol/L
Description: The number of participants who achieved a mean serum phosphorus value ≥ 1.13 and ≤ 1.78 mmol/L (3.5 to 5.5 mg/dL) during the effectiveness assessment phase.
Time Frame: Weeks 17 to 23
Population: All participants who received cinacalcet
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 71
Participants | 38
Statistical Analysis 1: Comparison: Cinacalcet; Test type: Superiority or Other; Percentage of participants = 53.5, 95% CI [41.9 to 65.1]

6. Secondary Outcome: Number of Participants Who Achieved a Mean CRP < 0.6 mg/dL
Description: The number of participants who achieved a mean C-reactive protein (CRP) level of < 0.6 mg/dL during the effectiveness assessment phase.
Time Frame: Weeks 17 to 23
Population: All participants who received cinacalcet
Measure: Number; unit: Participants
Arm/Group | Cinacalcet
Number analyzed (Participants) | 71
Participants | 33
Statistical Analysis 1: Comparison: Cinacalcet; Test type: Superiority or Other; Percentage of participants = 46.5, 95% CI [34.9 to 58.1]

ADVERSE EVENTS:
Time Frame: 23 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Cinacalcet
Serious Adverse Events (participants affected / at risk) | 27/71
Other Adverse Events (participants affected / at risk) | 42/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=71)
Acute Coronary Syndrome (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 5
Umbilical Hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Arteriovenous Fistula Site Infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Ross River Virus Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Arteriovenous Fistula Site Complication (Injury, poisoning and procedural complications) | 2
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 1
Complications of Transplanted Kidney (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Thrombosis in Device (Injury, poisoning and procedural complications) | 1
Blood Test Abnormal (Investigations) | 1
Platelet Count Decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hepatic Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Colic (Renal and urinary disorders) | 1
Renal Failure Chronic (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 1
Arteriovenous Fistula Operation (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 1
Iliac Artery Stenosis (Vascular disorders) | 1
Necrosis Ischaemic (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cinacalcet (N=71)
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 14
Nausea (Gastrointestinal disorders) | 18
Vomiting (Gastrointestinal disorders) | 14
Chest Pain (General disorders) | 5
Lower Respiratory Tract Infection (Infections and infestations) | 4
Anorexia (Metabolism and nutrition disorders) | 4
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 5
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4
Headache (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.